CLINICAL TRIAL: NCT07201818
Title: A Randomized Sham-Controlled Trial of Lymphatic Enhancement Technology in the Treatment of Fibromyalgia
Brief Title: LET for Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Arcturus Star Products (Unknown)
Responsible Party: Principal Investigator, Jason Zafereo, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU20251385
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia
Keywords: Lymphatic enhancement technology (LET); Chronic pain; Fibromyalgia; Autonomic Nervous System; Quantitative Sensory Testing
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: When it is determined that subjects are eligible for the study, the participants will be assigned by chance (like flipping a coin) to one of 2 study groups. Group 1 will receive active/real LET treatment, while group 2 will receive placebo/sham LET treatment.
Who Masked: Participant
Masking Description: Subjects will not know whether they are receiving the real or placebo treatment, but the researchers performing the treatment will know.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active LET group (Experimental): Participants in the active/real LET group will be treated with a machine that emits lights, sounds, and electrostatic energy. Three additional treatments will be administered over three weeks.
  Interventions: Device: Lymphatic Enhancement Technology (LET)
- Sham LET group (Sham Comparator): Participants in the placebo/sham LET group will be treated with a machine that emits lights and sounds, but no electrostatic energy. Three additional treatments will be administered over three weeks.
  Interventions: Device: Sham Lymphatic Enhancement Technology (LET)

INTERVENTIONS:
Device: Lymphatic Enhancement Technology (LET) — Lymphatic Enhancement Technology (LET) is an FDA-approved electrotherapeutic modality, with indications for addressing local lymphatic and vascular circulation as well as muscle pain and spasm. The Aria LET Elite Instrument (Arcturus Star, Cortez, Colorado) will be utilized for the intervention group.
  Arms: Active LET group
Device: Sham Lymphatic Enhancement Technology (LET) — A separate modified Aria Elite LET Instrument (Arcturus Star, Cortez, Colorado) will be utilized for the sham group. The sham LET device used for the control group will emit a light and sound similar to the true LET device, but will not emit energy waves.
  Arms: Sham LET group

SUMMARY:
The study is a double blinded, randomized, sham-controlled, parallel group trial conducted at UT Southwestern (UTSW) Medical Center. The purpose of this research study is to determine the effectiveness of Lymphatic Enhancement Technology (LET) treatment in patients with fibromyalgia. Participants will complete assessments of heart rate and blood pressure, pain thresholds to mechanical stimuli, and completion of quality-of-life surveys. In addition, participants will receive four treatments, one time per week, with either an active or sham LET device. Each visit will take between 45 minutes to 2 hours. A follow-up phone call or email from the study team will occur at 4 weeks after completion of the LET treatment. Total study duration is two months.

DETAILED DESCRIPTION:
At enrollment, participants will complete a baseline assessment including collection of demographic information (age, race/ethnicity, BMI, employment status, duration of symptoms, smoking history), past/current medical history, and current medications. The primary outcome measure of severity and functional impact of fibromyalgia symptoms will be collected using the Fibromyalgia Impact Questionnaire Revised (FIQR) at baseline, at each of the four treatment sessions, and one month after the last treatment. The following secondary outcome measures will be collected at baseline, immediately after the first treatment session, and before and after the fourth treatment session: 1. Pressure pain threshold (PPT), 2. temporal summation (TS) to pin prick, and 3. Autonomic cardiovascular function and conditioned pain modulation (CPM) during cold pressor test (CPT). Thirty-six participants will be randomized at the baseline testing session to receive 4 weekly treatments of active (n=18) or sham (n=18) LET. Opaque, sealed envelopes containing equal quantities of the number "1" or "2" will be placed into a container. On the first day of the study, participants will select an envelope that will only be opened by the treating clinician. The number "1" will designate participants to the active LET group, with the number "2" designating to the sham LET group. The treating clinician will record the participant's group assignment in order to administer the correct treatment throughout the study. The Aria LET Elite Instrument (Arcturus Star, Cortez, Colorado) will be utilized for the intervention and sham groups. The active device has two treatment wands that emit electrostatic energy, and give off a perceptible light and sound when they come in contact with the skin of the participant. The sham LET device used for the control group will also use two wands that emit a light and sound similar to the active LET device, but will not emit electrostatic energy waves. The device intensity ranges from 0-10 units which correlates to an amplitude of 12.9-38.25 microamps. Frequency ranges from 0-1000 units with a nonlinear correlation between 41-260 Hz. In the active treatment group, for session 1, the machine's intensity will be set to 3 units and a frequency of 300 units. For treatment session 2, the intensity and frequency will increase as tolerated to 4 units and 400 units, respectively. For treatment session 3, the intensity and frequency will increase as tolerated to 5 units and 500 units, respectively. For treatment session 4, the intensity and frequency will increase as tolerated to 6 units and 600 units, respectively. In the unlikely event that participants report an increase in fibromyalgia-related symptoms for more than two days after a treatment session, the treating clinicians will maintain (not increase) the intensity and frequency settings between visits. The treatment will utilize both wands contacting the skin of the participant and will progress in this treatment landmark order: terminus, jugulodigastric, parotid glands/sinuses, axilla, abdominal region, inguinal, lower/upper back. The clinicians will spend about 3 minutes on each landmark, spending more time in areas that exhibit more soft tissue resistance (detected through the wand), but staying within a total treatment time of 25 minutes. The control group will receive treatment using the same parameters, landmark progression, and treatment time on the sham device. All treatment parameters and participants' responses to treatment (treatment effect) will be documented at each visit. Additional measures will include a Blinding Fidelity Question administered at the end of the first and fourth treatment visit.

Using fibromyalgia as a target condition, the following aims will be tested:

1. Evaluate within- and between- group changes in severity and functional impact of fibromyalgia symptoms using the Fibromyalgia Impact Questionnaire-Revised (FIQR)
2. Evaluate within- and between- group changes in quantitative sensory testing (QST) and autonomic cardiovascular testing (ACT).
3. Correlate FIQR to QST and ACT values.

ELIGIBILITY:
Inclusion Criteria:

* meeting the American College of Rheumatology 2016 diagnostic criteria for fibromyalgia,
* female sex,
* ages 18-65 years,
* never received LET treatment,
* an FIQ score ≥39 (moderate severity), and
* no medication changes within 14 days prior to the start of the study or for the duration of the study.

Exclusion Criteria:

* currently receiving any other form of mind-body or exercise treatment,
* active blood clots,
* unexplained calf pain with concern for DVT,
* active infection,
* congestive heart failure,
* presence of an implanted pacemaker,
* pregnant or may be pregnant,
* active cancer or receiving cancer treatment, and
* having received any steroid injections within past 3 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in severity and functional impact of fibromyalgia symptoms as measured by FIQR at week 2 from baseline | Baseline, Week 2 pre-treatment
  The Revised Fibromyalgia Impact Questionnaire (FIQR) measures pain intensity and assesses how symptoms, including pain, interfere with a person's life. It is a 21-item, self-report questionnaire designed to evaluate the impact of fibromyalgia over the last seven days. The FIQR's assessment of pain intensity and interference is found within its three domains: Symptoms, Function and Overall Impact. By combining scores from these domains, the FIQR provides a comprehensive picture of how fibromyalgia symptoms, including pain intensity and interference, affect a patient's overall well-being. All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'.
Change in severity and functional impact of fibromyalgia symptoms as measured by FIQR at week 3 from baseline | Baseline, Week 3 pre-treatment
  The Revised Fibromyalgia Impact Questionnaire (FIQR) measures pain intensity and assesses how symptoms, including pain, interfere with a person's life. It is a 21-item, self-report questionnaire designed to evaluate the impact of fibromyalgia over the last seven days. The FIQR's assessment of pain intensity and interference is found within its three domains: Symptoms, Function and Overall Impact. By combining scores from these domains, the FIQR provides a comprehensive picture of how fibromyalgia symptoms, including pain intensity and interference, affect a patient's overall well-being. All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'.
Change in severity and functional impact of fibromyalgia symptoms as measured by FIQR at week 4 from baseline | Baseline, Week 4 pre-treatment
  The Revised Fibromyalgia Impact Questionnaire (FIQR) measures pain intensity and assesses how symptoms, including pain, interfere with a person's life. It is a 21-item, self-report questionnaire designed to evaluate the impact of fibromyalgia over the last seven days. The FIQR's assessment of pain intensity and interference is found within its three domains: Symptoms, Function and Overall Impact. By combining scores from these domains, the FIQR provides a comprehensive picture of how fibromyalgia symptoms, including pain intensity and interference, affect a patient's overall well-being. All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'.
Change in severity and functional impact of fibromyalgia symptoms as measured by FIQR at week 8 from baseline | Baseline, Week 8
  The Revised Fibromyalgia Impact Questionnaire (FIQR) measures pain intensity and assesses how symptoms, including pain, interfere with a person's life. It is a 21-item, self-report questionnaire designed to evaluate the impact of fibromyalgia over the last seven days. The FIQR's assessment of pain intensity and interference is found within its three domains: Symptoms, Function and Overall Impact. By combining scores from these domains, the FIQR provides a comprehensive picture of how fibromyalgia symptoms, including pain intensity and interference, affect a patient's overall well-being. All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'.

SECONDARY OUTCOMES:
Change quantitative sensory testing (QST) as assessed by PPT immediately after treatment 1 | Baseline, week 1 post treatment
  A pressure pain threshold (PPT) PPT measurements will be taken with a hand-held Algomed algometer mounted with a 1-cm2 probe and calibrated in kilopascals. Pressure will be applied at a constant rate of 30 kPa/s to two different locations bilaterally:1) Upper trapezius muscle at midway point between the C7 spinous process and acromion; 2) Gluteal muscles at midway point between PSIS and greater trochanter. Three measurements will be taken at each site and averaged to determine the final value for that site. Measurements will be expressed in kPa with a range of 0-800. Lower scores indicate more severe impact.
Change in quantitative sensory testing (QST) as assessed by PPT immediately after treatment 4 | Week 4 pre-treatment, week 4 post-treatment
  A pressure pain threshold (PPT) PPT measurements will be taken with a hand-held Algomed algometer mounted with a 1-cm2 probe and calibrated in kilopascals. Pressure will be applied at a constant rate of 30 kPa/s to two different locations bilaterally:1) Upper trapezius muscle at midway point between the C7 spinous process and acromion; 2) Gluteal muscles at midway point between PSIS and greater trochanter. Three measurements will be taken at each site and averaged to determine the final value for that site. Measurements will be expressed in kPa with a range of 0-800. Lower scores indicate more severe impact.
Change in quantitative sensory testing (QST) as assessed by PPT at week 4 post treatment from baseline | Baseline, week 4 post- treatment
  A pressure pain threshold (PPT) PPT measurements will be taken with a hand-held Algomed algometer mounted with a 1-cm2 probe and calibrated in kilopascals. Pressure will be applied at a constant rate of 30 kPa/s to two different locations bilaterally:1) Upper trapezius muscle at midway point between the C7 spinous process and acromion; 2) Gluteal muscles at midway point between PSIS and greater trochanter. Three measurements will be taken at each site and averaged to determine the final value for that site. Measurements will be expressed in kPa with a range of 0-800. Lower scores indicate more severe impact.
Change in quantitative sensory testing (QST) as assessed by temporal summation (TS) to pin prick immediately after treatment 1 | Baseline, week 1 post treatment
  A pin prick stimulator will be used to assess for TS at the same testing sites used for PPT. Subjects will first be exposed to a single stimulus, and then to 10 repetitive stimuli with an inter-stimulus interval (ISI) of 1 second applied within an area 1cm in diameter. Participants will be asked to rate the level of pinprick pain intensity using a numeric pain rating from 0-10 for the single stimulus, and then for the peak pain of the train of 10 stimuli. Two rounds of testing will be performed, and an average of the values will be calculated to obtain a single value for the single stimulus and the peak stimulus of the train. The ratio of the peak stimulus of the train to the single stimulus pain score will be calculated and used for analysis. Scores range from 0-10. Higher scores indicate more severe impact. Subjects will also report whether any aftersensations are present at either 15 or 30 seconds after each of the two trials.
Change in quantitative sensory testing (QST) as assessed by temporal summation (TS) to pin prick immediately after treatment 4 | Week 4 pre-treatment, week 4 post-treatment
  A pin prick stimulator will be used to assess for TS at the same testing sites used for PPT. Subjects will first be exposed to a single stimulus, and then to 10 repetitive stimuli with an inter-stimulus interval (ISI) of 1 second applied within an area 1cm in diameter. Participants will be asked to rate the level of pinprick pain intensity using a numeric pain rating from 0-10 for the single stimulus, and then for the peak pain of the train of 10 stimuli. Two rounds of testing will be performed, and an average of the values will be calculated to obtain a single value for the single stimulus and the peak stimulus of the train. The ratio of the peak stimulus of the train to the single stimulus pain score will be calculated and used for analysis. Scores range from 0-10. Higher scores indicate more severe impact. Subjects will also report whether any aftersensations are present at either 15 or 30 seconds after each of the two trials.
Change in quantitative sensory testing (QST) as assessed by temporal summation (TS) to pin prick at week 4 post treatment from baseline | Baseline, week 4 post treatment
  A pin prick stimulator will be used to assess for TS at the same testing sites used for PPT. Subjects will first be exposed to a single stimulus, and then to 10 repetitive stimuli with an inter-stimulus interval (ISI) of 1 second applied within an area 1cm in diameter. Participants will be asked to rate the level of pinprick pain intensity using a numeric pain rating from 0-10 for the single stimulus, and then for the peak pain of the train of 10 stimuli. Two rounds of testing will be performed, and an average of the values will be calculated to obtain a single value for the single stimulus and the peak stimulus of the train. The ratio of the peak stimulus of the train to the single stimulus pain score will be calculated and used for analysis. Scores range from 0-10. Higher scores indicate more severe impact. Subjects will also report whether any aftersensations are present at either 15 or 30 seconds after each of the two trials.
Change in quantitative sensory testing (QST) as assessed by CPM score immediately after treatment 1 | Baseline, week 1 post treatment
  Conditioned pain modulation (CPM) will be assessed via a PPT test stimulus applied to the upper trapezius for three trials. The average of the three PPT trials at the upper trapezius collected during the conditioning stimulus will be subtracted from the average of the three PPT trials collected before the CPT. Measurements of PPT will be expressed in kPa with a range of 0-800. Lower scores on CPM indicate more severe impact
Change in quantitative sensory testing (QST) as assessed by CPM score immediately after treatment 4 | Week 4 pre treatment, week 4 post treatment
  Conditioned pain modulation (CPM) will be assessed via a PPT test stimulus applied to the upper trapezius for three trials. The average of the three PPT trials at the upper trapezius collected during the conditioning stimulus will be subtracted from the average of the three PPT trials collected before the CPT. Measurements of PPT will be expressed in kPa with a range of 0-800. Lower scores on CPM indicate more severe impact
Change in quantitative sensory testing (QST) as assessed by CPM score at week 4 post treatment from baseline | Baseline, week 4 post treatment
  Conditioned pain modulation (CPM) will be assessed via a PPT test stimulus applied to the upper trapezius for three trials. The average of the three PPT trials at the upper trapezius collected during the conditioning stimulus will be subtracted from the average of the three PPT trials collected before the CPT. Measurements of PPT will be expressed in kPa with a range of 0-800. Lower scores on CPM indicate more severe impact
Change in autonomic cardiovascular testing (ACT) as assessed by Heart rate change during cold pressor task (CPT) immediately after treatment 1 | Baseline, week 1 post treatment
  Autonomic cardiovascular function measures of interest will include heart rate collected during the two conditions (before and during CPT). Measurements of HR will be expressed in BPM with a range of 0-200. Cardiovascular and sympathetic responses during each CPT will be calculated by subtracting the HR values collected during the 2nd minute of the CPT from the values collected during the rest period before the CPT. Lower scores on CPT indicate more severe impact.
Change in autonomic cardiovascular testing (ACT) as assessed by Heart rate change during cold pressor task (CPT) immediately after treatment 4 | Week 4 pre treatment, week 4 post treatment
  Autonomic cardiovascular function measures of interest will include heart rate collected during the two conditions (before and during CPT). Measurements of HR will be expressed in BPM with a range of 0-200.Cardiovascular and sympathetic responses during each CPT will be calculated by subtracting the HR values collected during the 2nd minute of the CPT from the values collected during the rest period before the CPT. Lower scores on CPT indicate more severe impact.
Change in autonomic cardiovascular testing (ACT) as assessed by Heart rate change during cold pressor task (CPT) at week 4 post treatment from baseline | Baseline, week 4 post treatment
  Autonomic cardiovascular function measures of interest will include heart rate collected during the two conditions (before and during CPT). Measurements of HR will be expressed in BPM with a range of 0-200.Cardiovascular and sympathetic responses during each CPT will be calculated by subtracting the HR values collected during the 2nd minute of the CPT from the values collected during the rest period before the CPT. Lower scores on CPT indicate more severe impact.
Change in autonomic cardiovascular testing (ACT) as assessed by change in systolic blood and diastolic pressure during cold pressor task (CPT) immediately after treatment 1 | Baseline, week 1 post treatment
  Autonomic cardiovascular function measures of interest will include blood pressure collected during the two conditions (before and during CPT). Measurements of blood pressure will be expressed in mmHg with a range of 0-200 for systolic and diastolic. Cardiovascular and sympathetic responses during each CPT will be calculated by subtracting the systolic and diastolic values collected during the 2nd minute of the CPT from the values collected during the rest period before the CPT. Lower scores on CPT indicate more severe impact.
Change in autonomic cardiovascular testing (ACT) as assessed by change in systolic blood and diastolic pressure during cold pressor task (CPT) immediately after treatment 4 | Week 4 pre treatment, week 4 post treatment
  Autonomic cardiovascular function measures of interest will include blood pressure collected during the two conditions (before and during CPT). Measurements of blood pressure will be expressed in mmHg with a range of 0-200 for systolic and diastolic. Cardiovascular and sympathetic responses during each CPT will be calculated by subtracting the systolic and diastolic values collected during the 2nd minute of the CPT from the values collected during the rest period before the CPT. Lower scores on CPT indicate more severe impact.
Change in autonomic cardiovascular testing (ACT) as assessed by change in systolic blood and diastolic pressure during cold pressor task (CPT) at week 4 post treatment from baseline | Baseline, week 4 post treatment
  Autonomic cardiovascular function measures of interest will include blood pressure collected during the two conditions (before and during CPT). Measurements of blood pressure will be expressed in mmHg with a range of 0-200 for systolic and diastolic. Cardiovascular and sympathetic responses during each CPT will be calculated by subtracting the systolic and diastolic values collected during the 2nd minute of the CPT from the values collected during the rest period before the CPT. Lower scores on CPT indicate more severe impact.

OTHER OUTCOMES:
Assessment of blinding fidelity immediately after treatment 1 | Week 1 post treatment
  Blinding fidelity will be assessed by asking the participants to indicate which group allocation they believe they are in after they have received treatment. Subjects may respond that they are in the experimental group, control group, or I don't know. Scores on the blinding index range from -1 to 1. A score of 0 indicated perfect blinding.
Assessment of blinding fidelity at week 4 post treatment | Week 4 post treatment
  Blinding fidelity will be assessed by asking the participants to indicate which group allocation they believe they are in after they have received treatment. Subjects may respond that they are in the experimental group, control group, or I don't know. Scores on the blinding index range from -1 to 1. A score of 0 indicated perfect blinding.
Treatment effect as assessed by change in pain intensity immediately after treatment 1 | Baseline, week 1 post treatment]
  Pain intensity will be assessed using the numeric pain rating scale (NPRS). Participants will be asked to rate their current level of pain on a scale from 0-10, with 0 representing no pain, and 10 their worst imaginable pain. Higher scores on NPRS indicate more severe impact.
Treatment effect as assessed by change in pain intensity immediately after treatment 2 | Week 2 pre treatment, week 2 post treatment
  Pain intensity will be assessed using the numeric pain rating scale (NPRS). Participants will be asked to rate their current level of pain on a scale from 0-10, with 0 representing no pain, and 10 their worst imaginable pain. Higher scores on NPRS indicate more severe impact.
Treatment effect as assessed by change in pain intensity immediately after treatment 3 | Week 3 pre treatment, week 3 post treatment
  Pain intensity will be assessed using the numeric pain rating scale (NPRS). Participants will be asked to rate their current level of pain on a scale from 0-10, with 0 representing no pain, and 10 their worst imaginable pain. Higher scores on NPRS indicate more severe impact.
Treatment effect as assessed by change in pain intensity immediately after treatment 4 | Week 4 pre treatment, week 4 post treatment
  Pain intensity will be assessed using the numeric pain rating scale (NPRS). Participants will be asked to rate their current level of pain on a scale from 0-10, with 0 representing no pain, and 10 their worst imaginable pain. Higher scores on NPRS indicate more severe impact.
Treatment effect as assessed by side effects reported after treatment 1 | Week 1 post treatment, Week 2 pre treatment
  Participants will be asked to report if they experienced any side effects during or after each treatment. Side effects may include experiencing a metallic taste or smell, increased bowel movements, increased fatigue or drowsiness, or increased fibromyalgia-related symptoms.
Treatment effect as assessed by side effects reported after treatment 2 | Week 2 post treatment, Week 3 pre treatment
  Participants will be asked to report if they experienced any side effects during or after each treatment. Side effects may include experiencing a metallic taste or smell, increased bowel movements, increased fatigue or drowsiness, or increased fibromyalgia-related symptoms.
Treatment effect as assessed by side effects reported after treatment 3 | Week 3 post treatment, Week 4 pre treatment
  Participants will be asked to report if they experienced any side effects during or after each treatment. Side effects may include experiencing a metallic taste or smell, increased bowel movements, increased fatigue or drowsiness, or increased fibromyalgia-related symptoms.
Treatment effect as assessed by side effects reported after treatment 4 | Week 4 post treatment, Week 8
  Participants will be asked to report if they experienced any side effects during or after each treatment. Side effects may include experiencing a metallic taste or smell, increased bowel movements, increased fatigue or drowsiness, or increased fibromyalgia-related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Zafereo, M.P.T, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center in the Allied Health Physical Therapy Clinic, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The data will be shared with Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. This data will be available for individual participant data meta-analysis. To gain access, data requestors will need to sign a data access agreement. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.
  Inquiries must be directed to Jason.Zafereo@UTSouthwestern.edu for requests for Information regarding submitting proposals and accessing data.